CLINICAL TRIAL: NCT03351062
Title: Multicenter Prospective, Parallel-controlled Phase III Clinical Study on Comparing Efficacy of Tamoxifen Versus Toremifene in CYP2D6 Intermediate/Poor Metabolizers of Premenopausal Patients With ER-positive Early Breast Cancer
Brief Title: Efficacy of Tamoxifen Versus Toremifene in CYP2D6 IM/PM of Premenopausal Patients With ER-positive Early Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Anti-Cancer Association (Other)
Collaborators: Fudan University (Other); Henan Cancer Hospital (Other Government); The First Hospital of Jilin University (Other); Southwest Hospital, China (Other); First Hospital of China Medical University (Other); Guangdong Provincial People's Hospital (Other); Harbin Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Jiangsu Provincial People's Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Zhejiang Cancer Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Union hospital of Fujian Medical University (Other); Hebei Tumor Hospital (Other); Hunan Cancer Hospital (Other); Affiliated Hospital of Qinghai University (Other); Wuhan TongJi Hospital (Other); Hainan People's Hospital (Other); The Third Affiliated Hospital of Kunming Medical College. (Other); The Third Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CYP2D6-1.1
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer Female
Keywords: premenopausal; early breast cancer; estrogen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen treatment group (Active Comparator): Patients in this group will receive tamoxifen treatment.
  Interventions: Drug: Tamoxifen
- Toremifene treatment group (Active Comparator): Patients in this group will receive Toremifene treatment.
  Interventions: Drug: Toremifene

INTERVENTIONS:
Drug: Tamoxifen — Patients will be given 10mg Tamoxifen twice a day.
  Other Names: Tamoxifen citrate
  Arms: Tamoxifen treatment group
Drug: Toremifene — Patients will be given 60mg Toremifene once a day.
  Other Names: fareston
  Arms: Toremifene treatment group

SUMMARY:
This clinical trial is designed to be a multi-center prospective, parallel-controlled Phase III clinical study. In this study, the efficacy of tamoxifen versus toremifene shall be compared in CYP2D6 intermediate/poor metabolizers of premenopausal patients with estrogen receptor-positive early breast cancer.

DETAILED DESCRIPTION:
STUDY BACKGROUND Breast cancer is a serious disease that threatens human health and life. Especially in China, the incidence rate is increasing year by year. According to WHO data, the incidence of breast cancer in China in 2020 will reach 214,000. Selective estrogen receptor modulators (SERMs) are a classic form of endocrine therapy for early breast cancers, but not all hormone receptor positive breast cancers benefit from specific SERMs. Numerous studies have shown that CYP2D6 variant carriers (around 50% CYP2D6 variant carriers in Chinese population) will not benefit a lot from tamoxifen, and combined use of CYP2D6 inhibitors will further affect the efficacy of tamoxifen. However, studies on another SERM drug - toremifene have shown that its metabolism and pharmacological effects are not influenced by CYP2D6 genotype or enzyme activity. Therefore, in the principle of individualized medicine, it is necessary to compare the efficacy of using tamoxifen and toremifene in CYP2D6 variant carriers in China so as to provide more guidance for clinical use.

OBJECTIVES:

1. The main purpose of this study is to compare 5-year disease-free survival rate of adjuvant endocrine therapy with tamoxifen and toremifene in premenopausal women with estrogen receptor-positive early breast cancer who are CYP2D6 intermediate/poor metabolizers.
2. The secondary purpose of this study includes:

   1. To compare 5-year overall survival (OS) and safety of adjuvant endocrine therapy with tamoxifen and toremifene in premenopausal patients with estrogen receptor-positive early breast cancer who are CYP2D6 intermediate/poor metabolizers.
   2. To compare the changes of plasma concentration of the parent drugs and metabolites of tamoxifen and toremifene in premenopausal patients with estrogen receptor-positive early breast cancer who are CYP2D6 intermediate/poor metabolizers.
   3. To assess the pharmacokinetics of tamoxifen and toremifene in premenopausal patients with estrogen receptor-positive early breast cancer who are CYP2D6 intermediate/poor metabolizers.

OUTLINE:

First, CYP2D6 genotype screening shall be conducted in premenopausal patients with estrogen receptor-positive early breast cancer in order to determine the frequency of different alleles. Then, patients who are CYP2D6 intermediate/poor metabolizers (with *4, *5, *10, *14, *17, *41 alleles) shall be stratified and randomized at the ratio of 1:1 ratio: allele status of CYP2D6 CYP2D6 intermediate/poor metabolizer (Heterozygous or homozygous), lymph node metastasis (with vs. without), prior chemotherapy (with vs. without), and HER2 status (positive vs. negative). Included patients shall be divided into two groups. One group will be given Tamoxifen (10mg Bid) for 5 years and the other group will be given toremifene (60mg qd) for 5 years. Then 5-year disease-free rate and overall survival and safety will be compared between these two groups. At Month 6, pharmacokinetic study on tamoxifen, toremifene and their metabolites will be conducted on patients.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women aged 18-50 years;
2. ECOG PS: 0-2 points;
3. Invasive breast cancer confirmed by histology with ER ≥ 10% (all test results should be reviewed and confirmed by Department of Pathology of the participant institution);
4. Participants have completed the standard local radical treatment (modified or conservative radical mastectomy) with or without neo-adjuvant/adjuvant chemotherapy or radiotherapy;
5. Participants must be able to understand this study and are willing to participate, agree to genotype screening and sign informed consent form with good compliance and cooperation in follow-ups;
6. Polymorphism analysis showed that patients are CYP2D6 * 4, * 5, * 10, * 14, * 17, * 41 allele carriers;
7. Hemoglobin ≥ 90g/L, neutrophils ≥ 1.5 × 109/L, platelets ≥ 75 × 109/L, AST and ALT ≤ 2.5 times the upper limit of normal (ULN), serum creatinine and urea nitrogen ≤ ULN.

Exclusion Criteria:

1. Patients have previously received neoadjuvant endocrine therapy or have started adjuvant endocrine therapy;
2. There are any comorbidities that may increase the level of sex hormones: such as pituitary adenomas, ovarian tumors, thymic carcinomas, etc.;
3. There are any comorbidities that may reduce the level of sex hormones such as hyperthyroidism, hypothyroidism, cirrhosis, severe malnutrition, Turner syndrome, lack of sex hormone synthetase, intracranial tumors, pituitary atrophy etc.;
4. Patients have undergone or planned to conduct ovariectomy or ovarian function inhibition;
5. Patients needs to take other medicines which can influence the activity of CYP2D6 (such as fluoxetine, paroxetine, quinidine, bupropion), CYP3A4 (such as erythromycin, acetylspiramycin, ritonavir, ketoconazole, nicardipine);
6. Patients have been treated with other trial medications in the past 2 weeks;
7. Pregnant or lactating women (women of childbearing age must have a negative pregnancy test within 14 days of the first dosing, and if pregnant, Patients are required for ultrasound examination to exclude pregnancy);
8. Women of childbearing age who are not willing to take effective contraception during treatment;
9. There are serious non-malignant tumor comorbidities that may affect long-term follow-up;
10. Patients have family history of endometrial, ovarian or other gynecologic malignancies;
11. Transvaginal ultrasound suggested more serious ovarian abnormalities or endometrial thickening;
12. Patients have had thrombotic events such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis, and pulmonary embolism within 6 months prior to study initiation;
13. Serious liver insufficiency with Child-Pugh C grade;
14. Serious cardiac insufficiency with New York Heart Association (NYHA) grade ≥III;
15. Patients are known severely allergic to study drug;
16. Patients have history of other malignancies in the past five years, except for cutaneous basal cell carcinoma and cervical carcinoma in situ which have been cured;
17. In other cases, the researchers don't think the subjects are suitable for participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 844 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | Within 5 years after randomization
  The time period from randomization to local or distant invasive cancer recurrence, contralateral invasive breast cancer, second (non-breast) primary invasive cancer and all-cause death

SECONDARY OUTCOMES:
Overall Survival | Within 5 years after randomization
  The time period from randomization to all-cause death
Adverse drug reaction | Within 5 years after administration
  The time period from administration to adverse events (dyslipidemia, endometrial hyperplasia) with confirmed, probably and possibly relevant relationship to trial medicine.
Serum drug concentration | Within 6 months after administration
  Blood level of trial medicines and their metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, Master, Principal Investigator — Fudan University
Locations (21):
- China (21):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Southwest Hospital, China, Chongqing, Chongqing Municipality
  - Union hospital of Fujian Medical University, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Hainan People's Hospital, Haikou, Hainan
  - Hebei Tumor Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Third Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - First Hospital of China Medical University, Shenyang, Lining
  - First Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The Third Affiliated Hospital of Kunming Medical College, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No